CLINICAL TRIAL: NCT03378687
Title: A Multi-center Clinical Study of Children With Status Epilepticus in China
Brief Title: A Clinical Study of Children With Status Epilepticus in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yi Wang, Vice President Chlidren's Hospital of Fudan University, Fudan University
Other Study IDs: 2016-165
Record Dates: First submitted 2017-05-15; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Status Epilepticus
Keywords: Status Epilepticus; Children; Multi-center; etiology; treatment; outcome; risk factor
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- status epileptius: Cases were patients 29 days to 18 years who were diagnosed with status epileptius in 35 hospitals in China between January 1， 2013 and December 31，2015.

SUMMARY:
Phase 1: The first part of study is a multi-center, retrospect study involving 38 hospitals. The program is a national epidemiological study on status epilepticus in Chinese children.The aims of the epidemiological study include:

1. to obtain national epidemiological data on the etiology, diagnosis,treatment,evaluation, risk factors , outcome and analyze the burden of disease.
2. to build a Collaborative Network in pediatric status epilepticus research.
3. to establish a national clinical database of pediatric status epilepticus.
4. to lay the foundation for the further prospective study.

Phase 2: The second part of study is a multi-center, prospective study involving 38 hospitals. The aim of the study is to set up guideline of Children with SE in China.

DETAILED DESCRIPTION:
Methods:

1. Case retrieval: The investigators query cases with a diagnostic code of SE via usage of the International Classification of Diseases, 10th revision (ICD-10) code G41.
2. Data collection:The subjects will be recruited from all hospitals.The investigators collect detailed information by a standardized questionnaire ,which contains each patient's age, gender, the date of occurrence of SE, past history of SE and seizures, etiology of SE, developmental history, underlying diseases, family history of seizures, duration of SE, seizure types of SE, laboratory data,EEG findings during SE and/or after SE, cranial CT and/or MRI findings after SE, medical treatment during the acute period and the outcome.The outcome include neurological sequelae, recurrence and death following SE.
3. The establishment of the database and data entry :The investigators established a database according the standardized questionnaire. Then the information will be put in the database by the responsible person of each hospital.
4. The standardized management of the database and quality control:There is a special person administrating the database and controlling the quality of data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnosis of Status Epilepticus(SE),which is defined as more than 30 minutes of either1).continuous seizure activity or 2).two or more sequential seizures without full recovery of consciousness between seizures, including Status Epilepticus (CSE) and Nonconvulsive Status Epilepticus(NCSE).
2. The age range: 29 days to <18years
3. Cases with complete clinical information.
4. Inpatient. All cases those meet full of the above 4 criterias are included in our study.

Exclusion Criteria:

1. A seizure less than 30 minutes
2. The newborn and more than 18 years old.

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients 29 days to 18years who were diagnosed with Status epilepticus in 34 hospitals between 1 January 2013 and 31 December 2015.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The outcome of children with SE at discharge | 2016.10.1-2017.6.30
  Use four measures to evaluate the outcome at discharge 1. Normal 2. With dysfunction 3. With secondary epilepsy 4. Death

SECONDARY OUTCOMES:
Glasgow Outcome Scale(GOS) | 2016.10.1-2017.6.30
  The GOS is a prognostic assessment tool for children with SE. GOS Score =1death GOS Score=2 Vegetative state ,Unable to interact with environment; unresponsive; GOS Score=3 Severe disability, Able to follow commands/ unable to live independently ;GOS Score=4 Moderate disability, Able to live independently; unable to return to work or school ;GOS Score=5 Good recovery，Able to return to work or school

CONTACTS AND LOCATIONS:
Overall Officials: Yi Wang, PhD,MD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Beijing Children's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- See also: The Children's Hospital of Fudan University (CHFU) is a service of the National Institute on Children. — http://ch.shmu.edu.cn/